CLINICAL TRIAL: NCT02684370
Title: BI 655066/ABBV-066 (Risankizumab) Versus Ustekinumab and Placebo Comparators in a Randomized Double Blind trIal for Maintenance Use in Moderate to Severe Plaque Type Psoriasis (UltIMMa-1)
Brief Title: BI 655066 (Risankizumab) Compared to Placebo and Active Comparator (Ustekinumab) in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M16-008; 2014-005117-23 (EudraCT Number); 1311.3 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-02-16; First posted 2016-02-18 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous; ustekinumab; Dermatologic Agents; ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous | interventions — risankizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Part A) (Placebo Comparator): Participants randomized to receive double-blind (DB) placebo by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: placebo for risankizumab; Drug: placebo for ustekinumab
- Ustekinumab (Part A) (Active Comparator): Participants randomized to receive double-blind (DB) ustekinumab 45 mg or 90 mg (based on screening weight) by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: placebo for risankizumab; Drug: ustekinumab
- Risankizumab (Part A) (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: risankizumab; Drug: placebo for ustekinumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Risankizumab (Part A)
Drug: placebo for risankizumab — Placebo for risankizumab administered by subcutaneous (SC) injection
  Arms: Placebo (Part A); Ustekinumab (Part A)
Drug: ustekinumab — Ustekinumab administered by subcutaneous (SC) injection
  Arms: Ustekinumab (Part A)
Drug: placebo for ustekinumab — Placebo for ustekinumab administered by subcutaneous (SC) injection
  Arms: Placebo (Part A); Risankizumab (Part A)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of BI 655066/ABBV-066 (risankizumab) for the treatment of moderate to severe chronic plaque psoriasis in adult patients.

DETAILED DESCRIPTION:
Participants were randomized to receive either placebo, ustekinumab, or risankizumab in Part A. All participants received 2 sets of injections to maintain the blind: the placebo arm received placebo for risankizumab and placebo for ustekinumab), the risankizumab arm received risankizumab and placebo for ustekinumab, and the ustekinumab arm received ustekinumab and placebo for risankizumab. Participants who received placebo in Part A switched to risankizumab in Part B; participants who received ustekinumab or risankizumab in Part A continued to receive the same treatment (ustekinumab or risankizumab) in Part B.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with age ≥18 years at screening.
* Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug.
* Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomisation):

  1. Have an involved body surface area (BSA) ≥10% and
  2. Have a Psoriasis Area and Severity Index (PASI) score ≥12 and
  3. Have a static Physician Global Assessment (sPGA) score of ≥3.
* Must be candidates for systemic therapy or phototherapy for psoriasis treatment, as assessed by the investigator.
* Must be a candidate for treatment with Stelara® (ustekinumab) according to local label.

Exclusion criteria:

* Patients with:

  1. non-plaque forms of psoriasis (including guttate, erythrodermic, or pustular)
  2. current drug-induced psoriasis (including an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
  3. active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis that might confound trial evaluations according to investigator's judgment
* Previous exposure to BI 655066.
* Previous exposure to ustekinumab (Stelara®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Background] Gordon KB, Strober B, Lebwohl M, Augustin M, Blauvelt A, Poulin Y, Papp KA, Sofen H, Puig L, Foley P, Ohtsuki M, Flack M, Geng Z, Gu Y, Valdes JM, Thompson EHZ, Bachelez H. Efficacy and safety of risankizumab in moderate-to-severe plaque psoriasis (UltIMMa-1 and UltIMMa-2): results from two double-blind, randomised, placebo-controlled and ustekinumab-controlled phase 3 trials. Lancet. 2018 Aug 25;392(10148):650-661. doi: 10.1016/S0140-6736(18)31713-6. Epub 2018 Aug 7. PMID 30097359
- [Derived] Strober B, Armstrong A, Rubant S, Patel M, Wu T, Photowala H, Crowley J. Switching to risankizumab from ustekinumab or adalimumab in plaque psoriasis patients improves PASI and DLQI outcomes for sub-optimal responders. J Dermatolog Treat. 2022 Nov;33(7):2991-2996. doi: 10.1080/09546634.2022.2095328. Epub 2022 Jul 31. PMID 35839335
- [Derived] Lebwohl MG, Soliman AM, Yang H, Wang J, Hagan K, Padilla B, Pinter A. Impact of Risankizumab on PASI90 and DLQI0/1 Duration in Moderate-to-Severe Psoriasis: A Post Hoc Analysis of Four Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Feb;12(2):407-418. doi: 10.1007/s13555-021-00660-3. Epub 2021 Dec 18. PMID 34921669
- [Derived] Augustin M, Lambert J, Zema C, Thompson EHZ, Yang M, Wu EQ, Garcia-Horton V, Geng Z, Valdes JM, Joshi A, Gordon KB. Effect of Risankizumab on Patient-Reported Outcomes in Moderate to Severe Psoriasis: The UltIMMa-1 and UltIMMa-2 Randomized Clinical Trials. JAMA Dermatol. 2020 Dec 1;156(12):1344-1353. doi: 10.1001/jamadermatol.2020.3617. PMID 33052382
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 560 subjects were enrolled; 54 subjects failed screening and are excluded from the analyses.
Groups:
- Placebo/Risankizumab (Part B): Participants randomized to receive placebo in Part A switched to risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Ustekinumab/Ustekinumab (Part B): Participants randomized to receive ustekinumab in Part A continued to receive ustekinumab 45 mg or 90 mg (based on screening weight) by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Risankizumab/Risankizumab (Part B): Participants randomized to receive risankizumab in Part A continued to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
Period: Part A
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Started (Intent-to-treat (ITT) population: All participants who were randomized at Week 0) | 102 | 100 | 304 | 0 | 0 | 0
Completed | 98 | 99 | 299 | 0 | 0 | 0
Not Completed | 4 | 1 | 5 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Withdrawal | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0
Period: Part B
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Started | 0 | 0 | 0 | 97 (1 participant who received placebo in Part A did not receive a dose of study drug in Part B) | 99 (Participants who received ustekinumab in Part A received ustekinumab in Part B) | 297 (2 participants who received risankizumab in Part A did not receive a dose of study drug in Part B)
Completed | 0 | 0 | 0 | 95 | 94 | 289
Not Completed | 0 | 0 | 0 | 2 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 5
Not completed — Subject Withdrawal | 0 | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All participants who were randomized at Week 0.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Total
Number analyzed (Participants) | 102 | 100 | 304 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13.63) | 46.5 (13.42) | 48.3 (13.39) | 48.1 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 92 | 145
  Male | 79 | 70 | 212 | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 23 | 47
  Not Hispanic or Latino | 90 | 88 | 281 | 459
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 7 | 11
  Asian | 28 | 22 | 86 | 136
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 1 | 1 | 10 | 12
  White | 71 | 74 | 200 | 345
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 4.9 | 75.3
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata (baseline weight [≤100 kg vs >100 kg] and prior exposure to tumor necrosis factor [TNF] antagonists [0 vs ≥1]). If there was a stratum containing zero count, 0.1 was added to each cell; adjusted difference in percentage = 70.3, 95% CI 2-sided [64.0 to 76.7] — 95% CI for adjusted difference of 2 treatment groups, calculated by Cochran-Mantel-Haenszel test adjusted for strata. If there was a stratum containing zero count, 0.1 was added to each cell

2. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 7.8 | 87.8
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata (baseline weight [≤100 kg vs >100 kg] and prior exposure to TNF antagonists [0 vs ≥1]). If there was a stratum containing zero count, 0.1 was added to each cell; adjusted difference in percentage = 79.9, 95% CI 2-sided [73.5 to 86.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 2.0 | 36.8
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 34.7, 95% CI 2-sided [28.6 to 40.8] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 0 | 35.9
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 35.5, 95% CI 2-sided [30.0 to 41.0] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 0 to 30, where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired.). A 5-point change from baseline is considered a clinically important difference. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 7.8 | 65.8
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 57.9, 95% CI 2-sided [50.4 to 65.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Achieving Psoriasis Symptoms Scale (PSS) Total Score of 0 at Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS total score is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. NRI was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 102 | 304
percentage of participants | 2.0 | 29.3
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 27.1, 95% CI 2-sided [21.2 to 32.9] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Achieving PASI90 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 1
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- Ustekinumab (Part A): Participants randomized to receive double-blind (DB) ustekinumab 45 mg or 90 mg (based on screening weight) SC at Weeks 0 and 4 (Part A).
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 42.0 | 75.3
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 33.5, 95% CI 2-sided [22.7 to 44.3] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 63.0 | 87.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 25.1, 95% CI 2-sided [15.2 to 35.0] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 4
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 12.0 | 35.9
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 23.8, 95% CI 2-sided [15.5 to 32.1] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 14.0 | 36.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 22.9, 95% CI 2-sided [14.3 to 31.6] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants Achieving PASI90 at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 1
Time Frame: Week 52
Population: ITT population. Non-responder imputation. Analysis performed on all participants randomized to ustekinumab or risankizumab treatment in Part A.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 100 | 304
percentage of participants | 44.0 | 81.9
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); P-value calculated according to the Cochran-Mantel-Haenszel test adjusted for baseline weight (≤100 kg vs >100 kg) and prior exposure to TNF antagonists (0 vs ≥1); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 38.3, 95% CI 2-sided [27.9 to 48.6] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 304 | 100
percentage of participants | 21.0 | 56.3
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata (baseline weight [≤100 kg vs >100 kg] and prior exposure to TNF] antagonists [0 vs ≥1]). If there was a stratum containing zero count, 0.1 was added to each cell; adjusted difference in percentage = 35.1, 95% CI 2-sided [25.7 to 44.6] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 52 in Participants Who Received Risankizumab Compared With Ustekinumab (Part B)
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
Number analyzed (Participants) | 100 | 304
percentage of participants | 21.0 | 57.6
Statistical Analysis 1: Comparison: Ustekinumab/Ustekinumab (Part B) vs Risankizumab/Risankizumab (Part B); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; adjusted difference in percentage = 36.5, 95% CI 2-sided [27.0 to 45.9] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 12 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 70.0 | 86.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; adjusted difference in percentage = 17.0, 95% CI 2-sided [7.4 to 26.6] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 12 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 2
Time Frame: Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 65.0 | 82.2
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; adjusted difference in percentage = 17.3, 95% CI 2-sided [7.3 to 27.3] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Percentage of Participants Achieving DLQI Score of 0 or 1 at Week 16 in Participants Who Received Risankizumab Compared With Ustekinumab (Part A)
Description: as for outcome 5
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 100 | 304
percentage of participants | 43.0 | 65.8
Statistical Analysis 1: Comparison: Ustekinumab (Part A) vs Risankizumab (Part A); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; adjusted difference in percentage = 23.0, 95% CI 2-sided [11.9 to 34.0] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: PSS Total Score: Change From Baseline to Week 16 in Participants Who Received Risankizumab Compared With Placebo (Part A)
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS total score is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. A negative change from Baseline indicates improvement. Last observation carried forward (LOCF) imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT population. Last observation carried forward. Participants randomized to placebo or risankizumab with an observed baseline PSS and at least one post-baseline PSS observation on or prior to Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 83 | 251
units on a scale | 0.157 (0.3476) | -5.608 (0.2254)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab (Part A); P-value calculated by the van Elteren test stratified for baseline weight (≤100 kg vs >100 kg) and prior exposure to TNF antagonists (0 vs ≥1); Test type: Other; p < 0.001, van Elteren test; Mean Difference (Final Values) = -5.765, 95% CI 2-sided [-6.496 to -5.035]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of study drug (up to 55 weeks).
Description: TEAEs and TESAEs in Part A are defined as events from the first dose of study drug in Part A until prior to the first dose in Part B (Week 16) or up to 105 days after the last dose of study drug if the participant discontinued in Part A; TEAEs and TESAEs in Part B are defined as events from the first dose of study drug in Part B (Week 16) until up to 105 days after the last dose of study drug.
Arm/Group | Placebo (Part A) | Ustekinumab (Part A) | Risankizumab (Part A) | Placebo/Risankizumab (Part B) | Ustekinumab/Ustekinumab (Part B) | Risankizumab/Risankizumab (Part B)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/100 | 0/304 | 0/97 | 0/99 | 0/297
Serious Adverse Events (participants affected / at risk) | 3/102 | 8/100 | 7/304 | 3/97 | 4/99 | 16/297
Other Adverse Events (participants affected / at risk) | 16/102 | 16/100 | 45/304 | 25/97 | 36/99 | 75/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=102) | Ustekinumab (Part A) (N=100) | Risankizumab (Part A) (N=304) | Placebo/Risankizumab (Part B) (N=97) | Ustekinumab/Ustekinumab (Part B) (N=99) | Risankizumab/Risankizumab (Part B) (N=297)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=102) | Ustekinumab (Part A) (N=100) | Risankizumab (Part A) (N=304) | Placebo/Risankizumab (Part B) (N=97) | Ustekinumab/Ustekinumab (Part B) (N=99) | Risankizumab/Risankizumab (Part B) (N=297)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 17 (20) | 8 (10) | 11 (14) | 30 (32)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 6 (7) | 6 (8) | 20 (24) | 15 (17) | 18 (20) | 40 (45)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 9 (9) | 3 (3) | 5 (5) | 5 (5)
Psoriasis (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.